CLINICAL TRIAL: NCT05749900
Title: First-line Trastuzumab Plus Chemoimmunotherapy for Biliary Tract Cancer (HERBOT Trial)
Brief Title: First-line Trastuzumab, Gemcitabine, Cisplatin and Nivolumab in Advanced HER2- Positive Biliary Tract Cancer: a Multicenter, Open-label, Single-arm Phase Ib/II Trial (HERBOT)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-1610
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: HER2 Positive Advanced/Metastatic/Nonresectable Biliary Tract Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab+Nivolumab+Gemcitabine+Cisplatin (Experimental): Trastuzumab+Nivolumab+Gemcitabine+Cisplatin
  Interventions: Drug: Trastuzumab+Nivolumab+Gemcitabine+Cisplatin

INTERVENTIONS:
Drug: Trastuzumab+Nivolumab+Gemcitabine+Cisplatin — Phase Ib Nivolumab 360mg IV q 3weeks Gemcitabine 1000mg/m2 IV D1, D8 q 3weeks Cisplatin 25mg/m2 IV D1, D8 q 3weeks Trastuzumab 8mg/kg (C1) then 6mg/kg IV q 3weeks Level -1 Nivolumab 360mg IV q 3weeks Gemcitabine 800mg/m2 IV D1, D8 q 3weeks Cisplatin 25mg/m2 IV D1, D8 q 3weeks Trastuzumab 8mg/kg (C1) then 6mg/kg IV q 3weeks

SUMMARY:
Biliary tract cancer is a rare malignant neoplasm including intrahepatic cholangiocarcinoma (IhCCA), extrahepatic cholangiocarcinoma (EhCCA) and Gallbladder cancer (GBC). Survival outcome of advanced BTCs are still poor and heterogeneity of tissue and molecular differences between BTCs limit the clinical studies in BTCs.

Combination therapy of Gemcitabine and Cisplatin has become the standard of care after the ABC-02 trial. This trial demonstrated that the addition of cisplatin to gemcitabine improved survival outcomes compared to that with gemcitabine alone. However, the median overall survival (OS) of Gem/Cis chemotherapy is only about one year.

Anti-Program cell death-1 (anti-PD-1) inhibitor monotherapy including Nivolumab (OPDIVO) had shown efficacy in refractory, advanced BTC. Various ICIs combined with Gem/Cis as the 1st line treatment in BTCs are under the trials. Combination of Nivolumab and Gem/Cis showed improved overall survival (15.4 months) in a small sized study (n=30) with tolerable side effects in advanced BTC patients. Recently reported interim analysis of phase III TOPAZ-1 trial (NCT03875235) showed Durvalumab, anti-PD-L1 agent, combined with Gem/Cis showed improvement of overall survival. Considering other studies currently ongoing, ICIs combined with Gem/Cis are thought to be the future standard of care in 1st line treatment of advanced stage BTCs.

HER2 amplification/overexpression is presented as many as 15% of total BTC patients. Basket trial of administration of pertuzumab and trastuzumab combination in previously treated HER2 positive advanced BTC patients showed promising overall response rate of 23%. Also, multicenter phase II study conducted by Korean investigators (KCSG-HB19-14) showed promising effect of Trastuzumab combined with modified FOLFOX in Gem/Cis refractory HER2 positive BTC patients with ORR of 29.4%. Moreover, preclinical data showed synergistic anti-cancer effect of trastuzumab combined with ICIs in HER2 positive cancers. Similar data are reported in HER2 positive gastric cancer that phase II and phase III clinical data showed 1st-line ICIs combined with trastuzumab and cytotoxic chemotherapy showed promising overall survival outcomes.

In treating HER2-positive advanced BTC, the triple combination of nivolumab, trastuzumab, and cytotoxic chemotherapy (Gem/Cis) may overcome innate resistance and activate an immune response to cancer along with inhibiting oncogenic signal from HER2 pathway, resulting in a synergistic effect with a longer response.

DETAILED DESCRIPTION:
This phase Ib/II study is designed to see whether trastuzumab+nivolumab+gemcitabine+cisplatin is active as palliative 1st line treatment for HER2-positive biliary tract cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically- or cytologically-confirmed biliary tract cancer (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gall bladder cancer)
2. HER2 positive biliary tract cancer (IHC 3+ or 2+ with ISH + (HER2/CEP17≥2.0) or ERBB2 gene copy number ≥ 6.0 by NGS)
3. Age (at the time of informed consent): 20 years and older
4. Previously untreated if unresectable/metastatic at initial diagnosis; or recurrent disease >6 months after curative surgery or adjuvant therapy (allow up to 1 cycle of gemcitabine-based chemotherapy for advanced/unresectable or metastatic cholangiocarcinoma prior to enrollment)
5. Explicit and voluntary consent to participate in the study obtained using a signed and dated informed consent form clearly and fully describing the purpose, potential risks, and any other critical issues regarding the study
6. Subject with measurable lesions according to RECIST v. 1.1
7. ECOG Performance Status Score 0 or 1
8. Patients with a life expectancy of at least 3 months
9. Patients whose latest laboratory data meet the below criteria within 14 days before enrollment.

   White blood cells ≥2,000/mm3 and neutrophils ≥1,500/mm3 Platelets ≥100,000/mm3 Hemoglobin ≥9.0 g/dL AST (GOT) and ALT (GPT) ≤3.0-fold the upper limit of normal (ULN) of the study site (or ≤5.0-fold the ULN of the study site in patients with liver metastases) Total bilirubin ≤1.5-fold the ULN of the study site Creatinine ≤1.5-fold the ULN of the study site or creatinine clearance (either the measured or estimated value using the Cockcroft-Gault equation) >45 mL/min INR ≤1.5-fold or prothrombin time ≤1.5-fold the ULN of the study site aPTT ≤1.5-fold the ULN of the study site
10. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons) #1 must agree to use contraception#2 from the time of informed consent until 5 months or more after the last dose of the investigational product. Also, women must agree not to breastfeed from the time of informed consent until 5 months or more after the last dose of the investigational product.
11. Men must agree to use contraception#2 from the start of study treatment until 7 months or more after the last dose of the investigational product.

    * 1. Women of childbearing potential are defined as all women after the onset of menstruation who are not postmenopausal and have not been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy). Postmenopause is defined as amenorrhea for ≥12 consecutive months without specific reasons. Women using oral contraceptives, intrauterine devices, or mechanical contraception such as contraceptive barriers are regarded as having childbearing potential.
    * 2. The subject must consent to use any of the following methods of contraception: vasectomy or condom for patients who are male or female subject's partner and tubal ligation, contraceptive diaphragm, intrauterine device, spermicide, or oral contraceptive for patients who are female or male subject's partner.
12. EF ≥ 50% via Transthoracic echocardiography or MUGA scan
13. Subjects willing to provide tumor biopsy tissue or excisional biopsy tissue.
14. Subjects with adequate organ function

Exclusion Criteria:

1. Patients treated with systemic chemotherapy, biologic therapy, immunotherapy, hormone therapy, or clinical trials for unresectable, locally advanced or metastatic biliary tract cancer. However, the following are excluded.

   1. If disease recurrence occurs 6 months after the last dose of adjuvant chemotherapy, previous adjuvant chemotherapy is permitted.
   2. 1 cycle of Gemcitabine-based anticancer therapy for locally advanced or metastatic cholangiocarcinoma prior to enrollment in this trial is permitted.
2. Patients with multiple primary cancers (with the exception of completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, or superficial bladder cancer, or any other cancer that has not recurred for at least 5 years)
3. Patients with residual adverse effects of prior therapy or effects of surgery that would affect the safety evaluation of the investigational product in the opinion of the investigator or sub-investigator.
4. Patients with current or past history of severe hypersensitivity to any other antibody products
5. Patients with concurrent autoimmune disease or history of chronic or recurrent autoimmune disease
6. Patients with a current or past history of interstitial lung disease or pulmonary fibrosis diagnosed based on imaging or clinical findings. Patients with radiation pneumonitis may be enrolled if the radiation pneumonitis has been confirmed as stable (beyond acute phase) without any concerns about recurrence.
7. Patients with concurrent diverticulitis or symptomatic gastrointestinal ulcerative disease
8. Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment. Patients may be enrolled if the metastasis is asymptomatic and requires no treatment.
9. Patients with pericardial fluid, pleural effusion, or ascites requiring treatment
10. Patients with uncontrollable, tumor-related pain
11. Patients who have experienced a transient ischemic attack or cerebrovascular accident within 180 days before enrollment
12. Patients with a history of uncontrollable or significant cardiovascular disease meeting any of the following criteria:

    1. Myocardial infarction within 180 days before enrollment
    2. Uncontrollable angina pectoris within 180 days before enrollment
    3. New York Heart Association (NYHA) Class III or IV congestive heart failure
    4. Uncontrollable hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥ 90 mmHg lasting 24 hours or more)
    5. Arrhythmia requiring treatment
13. Patients with uncontrollable diabetes mellitus
14. Patients with systemic infections requiring treatment (infection controlled by oral antibiotics is permitted)
15. Patients who have received systemic corticosteroids (prednisolone or equivalent > 10mg/day) (except for temporary use, e.g., for examination or prophylaxis of allergic reactions) or immunosuppressants within 28 days before enrollment
16. Patients who have received antineoplastic drugs (e.g., chemotherapy agents, molecular-targeted therapy agents, or immunotherapy agents) within 28 days before enrollment
17. Patients who have undergone surgical adhesion of the pleura or pericardium within 28 days before enrollment
18. Patients who have undergone surgery under general anesthesia within 28 days before enrollment
19. Patients who have undergone surgery involving local or topical anesthesia within 14 days before enrollment
20. Patients who have received radiotherapy within 28 days before enrollment, or radiotherapy to bone metastases within 14 days before enrollment
21. Patients who have received any radiopharmaceuticals (except for examination or diagnostic use of radiopharmaceuticals) within 56 days before enrollment
22. Patients with a positive test result for any of the following: HIV-1 antibody, HIV-2 antibody, HTLV-1 antibody, HBs antigen, or HCV antibody
23. Patients with active hepatitis B or C virus (Hepatitis patients can enrolled if HBV DNA and HCV RNA are controlled to less than 500 and are receiving stable antiviral treatment.)
24. Women who are pregnant or breastfeeding, or possibly pregnant
25. Patients who have received any other unapproved drug (e.g., investigational use of drugs, unapproved combined formulations, or unapproved dosage forms) within 28 days before enrollment
26. Patients who have previously received Nivolumab, anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CD137 antibody, anti-CTLA-4 antibody or other therapeutic antibodies or pharmacotherapies for regulation of T-cells
27. Patients judged to be incapable of providing consent for reasons such as concurrent dementia
28. Other patients judged by the investigator or sub-investigator to be inappropriate as subjects of this study
29. Patient with current or past history of hypersensitivity to Nivolumab.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Recommended Phase II Dose | up to 4 years
  Phase Ib: Recommended Phase II Dose decided during DLT periods
Phase II: Objective response rate, ORR | up to 4 years
  Phase II: Objective response rate, ORR: rate of patients with complete remission (CR) or partial remission (PR) based on RESIST1.1.

SECONDARY OUTCOMES:
Progression Free Survival, PFS | up to 4 years
  PFS is defined as time interval from cycle 1 day 1 to tumor progression/death/last follow-up
Overall Survival, OS | up to 4 years
  OS is defined as time interval from cycle 1 day 1 to tumor death/last follow-up.
Disease Control Rate, DCR | up to 4 years
  DCR is rate of patients with CR, PR, or SD per RECIST 1.1.
Duration of Response, DOR | up to 4 years
  DOR is defined as time interval from first response per RECIST 1.1 to tumor progression/death/last follow-up
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 4 years
  Safety per NCI CTCAE v5.0 ()Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 )
Quality of Life (QoL) | up to 4 years
  QoL determined by EORTC QLQ-C30 (QoL determined by EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Choong-kun Lee, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No